CLINICAL TRIAL: NCT04035694
Title: Web-based High School Media Literacy for Healthy Relationships
Brief Title: Evaluation Study of the Online High School Media Aware Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iRT-Media Aware HS-Phase II
Record Dates: First submitted 2019-07-16; First posted 2019-07-29 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-03

CONDITIONS: Sexual Behavior
Keywords: Adolescent sexual health; Media literacy education; Web-based programming
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive access to Media Aware.
  Interventions: Other: Media Aware Sexual Health - High School
- Delayed-Intervention Control (No Intervention): Participants will receive their regular health education programming not related to sexual health education or media literacy education.

INTERVENTIONS:
Other: Media Aware Sexual Health - High School — Media Aware is an online media literacy and sexual health education program developed for high school students that addresses the influence of media on sexual behaviors explicitly using established message processing theory. The program consists of 4 self-paced modules each with two to three lessons. Broadly, the modules cover healthy and unhealthy relationships, sexually transmitted infections, consent, substance use, pregnancy, protection and contraception, and communication between adolescents and their partners, parents, or health providers. Users also learn media literacy skills including message deconstruction to help examine the truth behind media messages.
  Other Names: Media Aware
  Arms: Intervention

SUMMARY:
The main aim of this study is to conduct a pretest-posttest RCT with a three-month follow-up to investigate the sustainability of outcomes in students who use the Media Aware program. Media Aware, a web-based media literacy education program for high school students to promote sexual and relationship health. Media Aware is designed to provide high school students with sexual health knowledge, media literacy skills, and the skills to make healthy decisions about sexual activity. This study will examine if behavioral indicators among students in the intervention group sustain, emerge, or diminish over time compared to students in the delayed intervention group.

ELIGIBILITY:
SCHOOL SITES:

Inclusion:

1. Schools must have students in 9th or 10th grade health education as this program is designed for use in these grades during health education classes.
2. Schools must agree to provide the Media Aware program during class periods as their sexual health education which means that an educator will facilitate the students taking the program.
3. Schools must have adequate technology for the students to use the web-based Media Aware program and complete the online questionnaires.
4. It must be feasible for iRT project staff members to travel to the school sites for the three data collection time points.

TEACHER PARTICIPANTS:

Inclusion:

1. Teacher's classrooms must have students in 9th or 10th grade as this program is designed for use in these grades.
2. Teachers must be able to ensure that participating students have computers and internet access during class periods as the program and questionnaires are web-based.

STUDENT PARTICIPANTS:

Inclusion:

1. Students must be in grades 9 or 10.
2. Students must be able to speak and read English because the study materials (e.g., questionnaires) are in English. However, parent permission and youth assent forms for the research study will be available in both English and Spanish.
3. Students must have appropriate parent permission to receive sexual health education per school districts' policy (i.e., opt-in policy or opt-out policy).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 590 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- innovation Research and Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All data collected will only be used for the research purposes in accordance with protocols approved by the IRB.

REFERENCES:
- [Background] Scull TM, Malik CV, Morrison A, Keefe EM. Study protocol for a randomized controlled trial to evaluate a web-based comprehensive sexual health and media literacy education program for high school students. Trials. 2020 Jan 8;21(1):50. doi: 10.1186/s13063-019-3992-1. PMID 31915060

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Delayed-Intervention Control
Started | 374 | 216
Completed | 374 | 216
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Delayed-Intervention Control | Total
Number analyzed (Participants) | 374 | 216 | 590
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.33 (.58) | 14.60 (.86) | 14.41 (.70)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 146 | 93 | 239
  Female | 197 | 96 | 293
  Nonbinary | 17 | 7 | 24
  Unknown or Not Reported | 14 | 20 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 27 | 72
  Not Hispanic or Latino | 313 | 167 | 480
  Unknown or Not Reported | 16 | 22 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 21 | 22 | 43
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 36 | 50 | 86
  White | 243 | 71 | 314
  More than one race | 51 | 43 | 94
  Unknown or Not Reported | 21 | 27 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 374 | 216 | 590
Sexual Experience [Count of Participants; unit: Participants] — Self-report of ever having oral, anal, or vaginal sex.
  Participants
    Yes | 40 | 35 | 75
    No | 280 | 137 | 417
    Unknown or Not Reported | 54 | 44 | 98
Academic Grades [Count of Participants; unit: Participants]
  Mostly As | 139 | 70 | 209
  As and Bs | 131 | 59 | 190
  Mostly Bs | 25 | 9 | 34
  Bs and Cs | 23 | 22 | 45
  Mostly Cs | 4 | 4 | 8
  Cs and Ds | 7 | 5 | 12
  Mostly Ds | 4 | 2 | 6
  Mostly Below Ds | 0 | 1 | 1
  Unknown or Not Reported | 41 | 44 | 85
Romantic Relationship Status [Count of Participants; unit: Participants]
  Yes | 55 | 39 | 94
  No/Unsure | 275 | 134 | 409
  Unknown or Not Reported | 44 | 43 | 87
Socioeconomic Status (SES) [Count of Participants; unit: Participants] — Self-report of eligibility for free or reduced lunch at school.
  Participants
    Yes | 43 | 71 | 114
    No/Unsure | 265 | 104 | 369
    Unknown or Not Reported | 66 | 41 | 107

OUTCOME MEASURES:

1. Primary Outcome: Willingness to Have Sex
Description: Participants are asked to indicate on a 4-point Likert scale (1=very unwilling; 2=unwilling; 3=willing; 4=very willing) how willing they are to have sex in a relationship context. (Imagine you were with a boyfriend/girlfriend and they say they love you. They want to have sex. In this situation, how willing would you be to have sex?).
Time Frame: posttest (approximately one week after pretest)
Population: The number of participants analyzed for this measure differs from the numbers in the Participant Flow module due to the fact that not all participants completed questionnaires at all time points and participants were able to skip questions on the questionnaire.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 244 | 122
units on a scale | 2.22 (.07) | 2.30 (.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — A series of multilevel regression models were estimated to determine the association between condition and each outcome, while controlling for the conditional non-independence of observations. Fixed effects included condition (intervention vs. control), the adolescent's pretest outcome score, and covariates (age, SES, race, sexual experience). The models included a random intercept for teacher and df were adjusted using the Satterthwaite adjustment; p = 0.41, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.08, Standard Error of Mean 0.08

2. Primary Outcome: Willingness to Have Sex
Description: as for outcome 1
Time Frame: follow-up (approximately three months after pretest)
Population: The number of participants analyzed for this measure differs from the numbers in the Participant Flow module due to the fact that not all participants completed questionnaires at all time points, participants were able to skip questions on the questionnaire. In addition, participants whose follow-up data were collected during the COVID-19 pandemic were excluded from the analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 190 | 56
units on a scale | 2.26 (0.08) | 2.42 (.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .11, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.16, Standard Error of Mean 0.10

3. Primary Outcome: Willingness to Engage in Unprotected Sex
Description: Participants are asked to indicate on a 4-point Likert scale (1=very unwilling; 2=unwilling; 3=willing; 4=very willing) how willing they are to engage in unprotected sex (Imagine you were with a boyfriend/girlfriend. They want to have sex, but neither of you have any form of protection. In this situation, how willing would you be to go ahead and have sex anyway?). (adapted from Gibbons, Gerrard, Blanton, & Russell, 2014)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 245 | 128
units on a scale | 1.69 (.07) | 1.75 (.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.54, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.06, Standard Error of Mean .09

4. Primary Outcome: Willingness to Engage in Unprotected Sex
Description: as for outcome 3
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 191 | 57
units on a scale | 1.72 (0.09) | 1.83 (0.12)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.38, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.12, Standard Error of Mean 0.11

5. Primary Outcome: Willingness to Hook up
Description: Participants are asked to indicate on a 4-point Likert scale (1=very unwilling; 2=unwilling; 3=willing; 4=very willing) how willing they are to have hook up even if they are not sure that they really want to (Imagine you were with a boyfriend/girlfriend. They want to hook-up, but you are not sure that you want to. In this situation, how willing would you be to go ahead and hook-up anyway?). (adapted from Gibbons, Gerrard, Blanton, & Russell, 2014)
Time Frame: posttest (approximately one week after pretest)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 244 | 128
units on a scale | 2.02 (.06) | 1.98 (.07)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.56, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = .04, Standard Error of Mean .07

6. Primary Outcome: Willingness to Hook up
Description: as for outcome 5
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 191 | 57
units on a scale | 1.98 (0.07) | 2.13 (0.09)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.09, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.14, Standard Error of Mean 0.08

7. Primary Outcome: Intentions to Engage in Sexual Activity With Another Person
Description: Participants are asked to indicate on a 4-point Likert scale (1=not at all likely; 2=unlikely; 3=likely; 4=extremely likely) how likely they are to engage in sexual activity in the next year (How likely is that you will have any type of sexual contact with another person (oral sex, anal sex, vaginal sex, or genital-to-genital contact) in the next year?). α = 0.77 (adapted from L'Engle, Brown, and Kenneavy, 2006)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 229 | 120
units on a scale | 2.03 (.07) | 1.96 (0.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.40, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.07, Standard Error of Mean 0.08

8. Primary Outcome: Intentions to Engage in Sexual Activity With Another Person
Description: as for outcome 7
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 184 | 57
units on a scale | 1.97 (0.09) | 2.00 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.74, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.03, Standard Error of Mean 0.09

9. Primary Outcome: Condom Use Intentions
Description: Participants are asked to indicate on a 4-point Likert scale (1=not at all likely; 2=unlikely; 3=likely; 4=extremely likely) how likely they are to use protection (if you were to have vaginal or anal sex, how likely would you be to use a condom?). (adapted from Jemmott and Jemmott, 1991)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 235 | 124
units on a scale | 3.46 (0.06) | 3.42 (0.07)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.66, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.03, Standard Error of Mean 0.07

10. Primary Outcome: Condom Use Intentions
Description: as for outcome 9
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 188 | 56
units on a scale | 3.53 (0.08) | 3.51 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.78, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.03, Standard Error of Mean 0.09

11. Primary Outcome: Birth Control Use Intentions (Other Than Condoms)
Description: Participants are asked to indicate on a 4-point Likert scale (1=not at all likely; 2=unlikely; 3=likely; 4=extremely likely) how likely they are to use protection (if you were to have vaginal sex, how likely would you be to use birth control other than condoms?). (adapted from Jemmott and Jemmott, 1991)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 235 | 123
units on a scale | 2.99 (0.11) | 2.89 (0.13)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.52, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.10, Standard Error of Mean 0.15

12. Primary Outcome: Birth Control Use Intentions (Other Than Condoms)
Description: as for outcome 11
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 185 | 57
units on a scale | 2.83 (0.12) | 2.76 (0.17)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.74, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.07, Standard Error of Mean 0.17

13. Primary Outcome: Protection Intentions During Oral Sex
Description: Participants are asked to indicate on a 4-point Likert scale (1=not at all likely; 2=unlikely; 3=likely; 4=extremely likely) how likely they are to use protection (if you were to decide to have oral sex, how likely would you be to use a condom or dental dam?). (adapted from Jemmott and Jemmott, 1991)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 236 | 124
units on a scale | 2.94 (0.10) | 2.77 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.21, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Median Difference (Net) = 0.17, Standard Error of Mean 0.13

14. Primary Outcome: Protection Intentions During Oral Sex
Description: as for outcome 13
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 186 | 57
units on a scale | 2.83 (0.11) | 2.68 (0.15)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.27, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.14, Standard Error of Mean 0.13

15. Secondary Outcome: Perceived Realism of Media Messages
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) the degree to which they agreed that teens on the media (e.g., Teens in the media do things that average teens do.). (adapted from Austin and Johnson, 1997, α=0.80)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 250 | 137
units on a scale | 2.02 (0.05) | 2.23 (0.06)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Median Difference (Net) = -0.21, Standard Error of Mean 0.07

16. Secondary Outcome: Perceived Realism of Media Messages
Description: as for outcome 15
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 217 | 59
units on a scale | 2.03 (0.08) | 2.19 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.23, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.15, Standard Error of Mean 0.11

17. Secondary Outcome: Acceptance of Dating Violence
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly 2=disagree; 3=disagree; 4=agree; strongly agree) their level of agreement on several items pertaining to dating violence (e.g., It is okay for people to hit their girlfriends/boyfriends if they did something to make them mad.). (adapted from Foshee, Bauman, Ennett, Suchindran, Benefield, and Linder, 2005 α=0.73)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 249 | 135
units on a scale | 1.40 (0.04) | 1.48 (0.04)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.09, Standard Error of Mean 0.05

18. Secondary Outcome: Acceptance of Dating Violence
Description: as for outcome 17
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 219 | 60
units on a scale | 1.36 (0.07) | 1.36 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.95, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.01, Standard Error of Mean 0.11

19. Secondary Outcome: Advertisement Deconstruction Skills
Description: Participants are shown an advertisement and asked to describe it in detail including noting marketing strategies and any missing information (e.g., How are advertisers trying to get someone to buy this product?). Qualitative responses to the questions are coded by trained project staff members once inter-coder reliability is established, and scores will be summed to create an overall deconstruction skills composite variable. (adapted from Kupersmidt, Scull, & Benson, 2012)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 250 | 131
units on a scale | 4.46 (0.52) | 3.47 (0.53)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.19, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.99, Standard Error of Mean 0.72

20. Secondary Outcome: Advertisement Deconstruction Skills
Description: Participants are shown an advertisement and asked to describe it in detail including noting marketing strategies and any missing information (e.g., How are advertisers trying to get someone to buy this product?). Qualitative responses to the questions are coded by trained project staff members once inter-coder reliability is established, and scores will be summed to create an overall deconstruction skills composite variable (adapted from Kupersmidt, Scull, & Benson, 2012).
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 223 | 60
units on a scale | 5.30 (0.35) | 5.37 (0.55)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.92, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.06, Standard Error of Mean 0.59

21. Secondary Outcome: Media Message Completeness
Description: Participants are shown an advertisement and asked to indicate on a 4-point Likert scale (1=incomplete to 4=complete) how complete the information included in an advertisement is (e.g., How complete is the information in this advertisement?).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 247 | 130
units on a scale | 2.17 (0.10) | 2.20 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.81, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Median Difference (Net) = -0.03, Standard Error of Mean 0.13

22. Secondary Outcome: Media Message Completeness
Description: as for outcome 21
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 217 | 58
units on a scale | 2.27 (0.11) | 2.23 (0.16)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.81, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.04, Standard Error of Mean 0.16

23. Secondary Outcome: Media Skepticism
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) the degree to which they agree with several statements about media (e.g., Media are dishonest about what happens if people have sex.). (adapted from Scull, Malik, and Kupersmidt, 2014, α=0.86)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 251 | 136
units on a scale | 2.93 (0.07) | 2.78 (0.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.14, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.15, Standard Error of Mean 0.10

24. Secondary Outcome: Media Skepticism
Description: as for outcome 23
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 218 | 60
units on a scale | 3.04 (0.09) | 3.01 (0.14)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.82, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.04, Standard Error of Mean 0.15

25. Secondary Outcome: Acceptance of Strict Gender Role Stereotypes
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) their level of agreement on several items pertaining to strict gender role stereotypes (e.g., Raising children is primarily a woman's responsibility.). (adapted from Foshee, Bauman, Ennett, Suchindran, Benefield, and Linder, 2005 α=0.87)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 252 | 136
units on a scale | 1.51 (0.04) | 1.52 (0.05)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.97, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Median Difference (Net) = 0.00, Standard Error of Mean 0.05

26. Secondary Outcome: Acceptance of Strict Gender Role Stereotypes
Description: as for outcome 25
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 219 | 60
units on a scale | 1.44 (0.06) | 1.45 (0.09)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.89, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.01, Standard Error of Mean 0.09

27. Secondary Outcome: Acceptance of Rape Myths
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) their level of agreement on several items pertaining to myths about rape (e.g., It shouldn't be considered rape if a guy is drunk and didn't realize what he was doing.). (adapted from Illinois Rape Myth Acceptance-Short Form (IRMA-SF; 7 pt. scale); Payne et al., (1999); McMahon & Farmer (2011), α=0.88)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 251 | 135
units on a scale | 1.35 (0.04) | 1.33 (0.04)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.69, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.02, Standard Error of Mean 0.05

28. Secondary Outcome: Acceptance of Rape Myths
Description: as for outcome 27
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 219 | 58
units on a scale | 1.31 (0.05) | 1.28 (0.07)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.63, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.03, Standard Error of Mean 0.06

29. Secondary Outcome: Intentions to Intervene as Bystander
Description: Participants are asked to indicate on a 4-point Likert scale (1=not likely at all; 2=Unlikely; 3=Likely; 4=Extremely likely) how likely they would be to intervene as a bystander (e.g., Approach a friend if I thought they were in an abusive relationship and let them know that I am here to help.). (adapted from Banyard, 2005)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 247 | 136
units on a scale | 3.10 (0.06) | 3.08 (0.06)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.79, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.02, Standard Error of Mean 0.07

30. Secondary Outcome: Intentions to Intervene as Bystander
Description: as for outcome 29
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 217 | 58
units on a scale | 3.13 (0.09) | 3.11 (0.15)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.93, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.02, Standard Error of Mean 0.16

31. Secondary Outcome: Efficacy to Intervene as Bystander
Description: Participants are asked to indicate on a scale of 0 (Can't do) to 100 (Very Certain) their degree of confidence in several behaviors (e.g., I could talk to a friend who I suspected is in an abusive relationship.). (adapted from Banyard, 2005)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 251 | 136
units on a scale | 74.26 (1.68) | 71.28 (1.85)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .20, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 2.98, Standard Error of Mean 2.18

32. Secondary Outcome: Efficacy to Intervene as Bystander
Description: as for outcome 31
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 217 | 57
units on a scale | 75.96 (1.90) | 70.97 (2.70)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.11, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 5.00, Standard Error of Mean 2.52

33. Secondary Outcome: Descriptive Norms Regarding Teen Sexual Activity
Description: Participants are asked to indicate what percentage [0% = no teens; 100% = all teens] of teens engage in sexual activity (e.g., oral sex, vaginal sex, anal sex). (adapted from Scull, Kupersmidt, Malik, and Keefe, 2018)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of teens sexually active
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 238 | 129
percentage of teens sexually active | 36.10 (1.85) | 43.02 (2.01)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -6.93, Standard Error of Mean 2.38

34. Secondary Outcome: Descriptive Norms Regarding Teen Sexual Activity
Description: as for outcome 33
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of teens sexually active
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 192 | 55
percentage of teens sexually active | 38.65 (2.67) | 40.89 (4.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.64, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -2.24, Standard Error of Mean 4.45

35. Secondary Outcome: Descriptive Norms Regarding Teen Risky Sexual Activity
Description: Participants are asked to indicate what percentage [0% = no teens; 100% = all teens] of teens engage in risky sexual activities (e.g., What percentage of teens have sex with someone who is much older?). (adapted from Scull, Kupersmidt, Malik, and Keefe, 2018)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of teens having risky sex
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 235 | 123
percentage of teens having risky sex | 30.89 (2.00) | 37.35 (2.18)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.03, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -6.46, Standard Error of Mean 2.53

36. Secondary Outcome: Descriptive Norms Regarding Teen Risky Sexual Activity
Description: as for outcome 35
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of teens having risky sex
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 190 | 51
percentage of teens having risky sex | 36.39 (2.19) | 35.17 (3.00)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.65, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 1.23, Standard Error of Mean 2.68

37. Secondary Outcome: Sexual Health Knowledge
Description: Participants are asked several multiple choice and True/False questions about sexual health (e.g., True or false: You can tell someone has an STI by looking at him/her.).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 236 | 124
score on a scale | 11.38 (0.13) | 10.72 (0.14)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < .01, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.65, Standard Error of Mean 0.15

38. Secondary Outcome: Sexual Health Knowledge
Description: as for outcome 37
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 207 | 56
score on a scale | 11.34 (0.18) | 11.06 (0.24)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.20, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.28, Standard Error of Mean 0.22

39. Secondary Outcome: Descriptive Norms Regarding Sexual Health Communication
Description: Participants are asked to indicate what percentage [0% = no teens; 100% = all teens] of teens communicate with parents, health providers, or another trusted adult (e.g., Before deciding to have sex, what percentage of teens talk with their boy/girlfriend about sexual health?). (adapted from Scull, Kupersmidt, Malik, and Keefe, 2018)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of teens communicating
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 236 | 123
percentage of teens communicating | 39.95 (1.88) | 37.16 (2.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.28, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 2.79, Standard Error of Mean 2.22

40. Secondary Outcome: Descriptive Norms Regarding Sexual Health Communication
Description: as for outcome 39
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of teens communicating
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 191 | 52
percentage of teens communicating | 40.97 (2.27) | 39.41 (3.15)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.58, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Median Difference (Net) = 1.56, Standard Error of Mean 2.77

41. Secondary Outcome: Efficacy to Negotiate Contraception/Protection Use
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) how effectively they could convince a partner to use contraception (e.g., If I decided to have sex, I could talk to any potential partner to make him/her understand why we should use condoms or other contraception.).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 239 | 131
units on a scale | 3.19 (0.08) | 3.11 (0.09)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.49, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.07, Standard Error of Mean 0.10

42. Secondary Outcome: Efficacy to Negotiate Contraception/Protection Use
Description: as for outcome 41
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 190 | 56
units on a scale | 3.30 (0.09) | 3.39 (0.13)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .55, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.09, Standard Error of Mean 0.14

43. Secondary Outcome: Efficacy to Use Contraception/Protection
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) how effectively they could get and use contraception (e.g., If I wanted to, I could get condoms or another form of contraception.).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 239 | 131
units on a scale | 3.06 (0.07) | 3.00 (0.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.54, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.06, Standard Error of Mean 0.09

44. Secondary Outcome: Efficacy to Use Contraception/Protection
Description: as for outcome 43
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 193 | 57
units on a scale | 3.22 (0.08) | 3.23 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.95, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.01, Standard Error of Mean 0.10

45. Secondary Outcome: Descriptive Norms Regarding Teen Birth Control Use
Description: Participants are asked to indicate what percentage [0% = no teens; 100% = all teens] of teens use contraception (e.g., What percentage of teens who have oral sex use a condom or a dental dam?). (adapted from Scull, Kupersmidt, Malik, and Keefe, 2018)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of teens using BC
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 238 | 121
percentage of teens using BC | 54.09 (1.86) | 58.34 (2.07)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Median Difference (Net) = -4.25, Standard Error of Mean 2.15

46. Secondary Outcome: Descriptive Norms Regarding Teen Birth Control Use
Description: as for outcome 45
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of teens using BC
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 190 | 50
percentage of teens using BC | 53.89 (2.64) | 52.52 (3.93)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.75, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 1.37, Standard Error of Mean 3.84

47. Secondary Outcome: Efficacy to Communicate Before Sex
Description: Participants are asked to indicate on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) how effectively they could communicate with others about sexual health (e.g., I could talk with a boy/girlfriend about using condoms for sexually transmitted infection protection.). (adapted from Scull, Malik, & Kupersmidt, 2014)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 240 | 131
units on a scale | 2.93 (0.07) | 2.79 (0.07)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.14, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.14, Standard Error of Mean 0.09

48. Secondary Outcome: Efficacy to Communicate Before Sex
Description: as for outcome 47
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 193 | 56
units on a scale | 2.92 (0.07) | 2.74 (0.09)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.03, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.18, Standard Error of Mean 0.08

49. Secondary Outcome: Intent to Communicate Before Sex
Description: Participants are asked to indicate on a 4-point Likert scale (1=not at all likely; 2=unlikely; 3=likely; 4=extremely likely) how likely they are to communicate with others before sexual activity (e.g., Before deciding to have sex, how likely would you be to talk with your parents or another trusted adult about sexual health?). (adapted from Scull, Malik, & Kupersmidt, 2014)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 237 | 128
units on a scale | 2.82 (0.06) | 2.64 (0.06)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.18, Standard Error of Mean 0.06

50. Secondary Outcome: Intent to Communicate Before Sex
Description: as for outcome 49
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 187 | 57
units on a scale | 2.80 (0.07) | 2.60 (0.09)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.02, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.20, Standard Error of Mean 0.08

51. Secondary Outcome: Cognitive Elaboration While Viewing an Advertisement
Description: Participants are shown an advertisement and asked to indicate on a 4-point Likert scale (1=not much at all; 2=a little; 3=a good amount; 4=a lot) the extent to which they: 1) thought about the ad; 2) spent time thinking about the ad; and 3) paid attention to the ad. (adapted from Shiv, Britton, and Payne, 2004)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 249 | 133
units on a scale | 2.01 (0.06) | 1.86 (0.06)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.03, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.14, Standard Error of Mean 0.06

52. Secondary Outcome: Cognitive Elaboration While Viewing an Advertisement
Description: as for outcome 51
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 217 | 59
units on a scale | 1.94 (0.09) | 2.02 (0.14)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.57, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.08, Standard Error of Mean 0.13

53. Secondary Outcome: Communication With a Doctor or Other Health Professional About Sexual Health
Description: Participants are asked on a 4-point Likert scale (1never; 2=rarely; 3=sometimes; 4=often) about their frequency of sexual health communication with a doctor or other health professional (e.g., How often do you talk with a doctor or other health professional about sexual health?).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 238 | 126
units on a scale | 1.98 (0.07) | 1.97 (0.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.91, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.01, Standard Error of Mean 0.08

54. Secondary Outcome: Communication With a Doctor or Other Health Professional About Sexual Health
Description: as for outcome 53
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 184 | 58
units on a scale | 1.83 (0.09) | 1.79 (0.12)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.72, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.04, Standard Error of Mean 0.11

55. Secondary Outcome: Communication With a Parent or Other Trusted Adult About Sexual Health
Description: Participants are asked on a 4-point Likert scale (1never; 2=rarely; 3=sometimes; 4=often) about their frequency of sexual health communication with a doctor or trusted adult (e.g., How often do you talk with a parent or other trusted professional about sexual health?).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 238 | 125
units on a scale | 2.15 (0.08) | 1.95 (0.09)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.07, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.20, Standard Error of Mean 0.09

56. Secondary Outcome: Communication With a Parent or Other Trusted Adult About Sexual Health
Description: as for outcome 55
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 184 | 58
units on a scale | 1.95 (0.09) | 2.00 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.56, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.06, Standard Error of Mean 0.10

57. Secondary Outcome: Communication With a Boyfriend or Girlfriend About Sexual Health
Description: Participants are asked on a 4-point Likert scale (1never; 2=rarely; 3=sometimes; 4=often) about their frequency of sexual health communication with a boyfriend/girlfriend (e.g., How often do you talk with your boyfriend/girlfriend about sexual health?).
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 222 | 120
units on a scale | 1.93 (0.09) | 1.77 (0.10)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.17, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.16, Standard Error of Mean 0.11

58. Secondary Outcome: Communication With a Boyfriend or Girlfriend About Sexual Health
Description: as for outcome 57
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 170 | 55
units on a scale | 1.95 (0.10) | 1.96 (0.13)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.89, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.02, Standard Error of Mean 0.12

59. Other Pre Specified Outcome: Counterarguing While Viewing an Advertisement
Description: Participants are shown an advertisement and asked to indicate on a 4-point Likert scale (1=not much at all; 2=a little; 3=a good amount; 4=a lot) the extent to which they: 1) wanted to argue back to what it was saying; 2) thought of ways they disagreed with what was presented; 3) thought of ways that the information being presented was inaccurate or misleading; and 4) found themselves looking for flaws in the way information was presented in the ad. (adapted from Moyer-Gusé and Nabi, 2010)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 248 | 133
units on a scale | 2.01 (0.07) | 1.90 (0.07)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .20, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = 0.11, Standard Error of Mean 0.08

60. Other Pre Specified Outcome: Counterarguing While Viewing an Advertisement
Description: as for outcome 59
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 216 | 59
units on a scale | 1.87 (0.10) | 1.92 (0.16)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.78, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.05, Standard Error of Mean 0.16

61. Other Pre Specified Outcome: Advertisement Credibility
Description: Participants are shown an advertisement and asked to indicate on a 4-point Likert scale (variable) how 1) believable; 2) truthful; 3) trustworthy they find the advertisement. (adapted from MacKenzie, Lutz, and Belch, 1986)
Time Frame: posttest (approximately one week after pretest)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 250 | 132
units on a scale | 2.12 (0.07) | 2.20 (0.08)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.41, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.08, Standard Error of Mean 0.09

62. Other Pre Specified Outcome: Advertisement Credibility
Description: as for outcome 61
Time Frame: follow-up (approximately three months after pretest)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Delayed-Intervention Control
Number analyzed (Participants) | 216 | 59
units on a scale | 2.01 (0.08) | 2.14 (0.12)
Statistical Analysis 1: Comparison: Intervention vs Delayed-Intervention Control; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.34, Mixed Models Analysis; The df were adjusted to take into account random effects using Satterthwaite df adjustment for mixed models; Mean Difference (Net) = -0.13, Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: Research staff members scanned the incoming online questionnaire data on a regularly basis and recorded any problems seen or concerns about any participants over the study timeframe (approx. 3 months).
Description: Study risks were defined as discomfort with assessment procedures/content, or breach of confidentiality. Measures were taken to provide confidentiality with respect to questionnaire responses and program process data. To minimize the risk of discomfort for participants, participants could skip any question and quit participation at any time. Research staff scanned the incoming data on a regularly basis to record any concerns about any participants. No adverse events were reported.
Arm/Group | Intervention | Delayed-Intervention Control
All-Cause Mortality (participants affected / at risk) | 0/374 | 0/216
Serious Adverse Events (participants affected / at risk) | 0/374 | 0/216
Other Adverse Events (participants affected / at risk) | 0/374 | 0/216

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic began during this trial, and primarily impacted the collection of follow-up data. Data collection procedures were revised to take into account social distancing measures and schools switching to remote learning. Response rates were lower and analyses revealed systematic differences between groups; therefore, data from these students were not included in the follow-up analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT04035694/Prot_SAP_000.pdf